CLINICAL TRIAL: NCT06951646
Title: ctDNA-MRD Guided Escalation of Ivonescimab and Docetaxel in Advanced NSCLC With Long-Term Responses to First-line Immunotherapy: a Randomized, Open-label, Phase II Trial (CR1STAL-Adaptive)
Brief Title: ctDNA-MRD Guided Escalation of Ivonescimab and Docetaxel in Advanced NSCLC With Long-Term Responses to First-line Immunotherapy (CR1STAL-Adaptive)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Akeso-Sino Pharma Co., Ltd. (Unknown); Nanjing Shihejiyin Technology, Inc. (Industry)
Responsible Party: Principal Investigator, Fang Wu, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYG20240091
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Immune Checkpoint Inhibitors (ICIs)
Keywords: Non Small Cell Lung Cancer (NSCLC); Immune Checkpoint Inhibitors (ICIs); Circulating-tumor DNA (ctDNA); Minimal Residual Disease (MRD); Ivonescimab (AK112); Adaptive Therapy; Bispecific Antibody; Escalation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to the standard treatment group or the advanced treatment group. In the event of disease progression (PD), they are optional to receive the Ivonescimab plus docetaxel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Other): For ctDNA-positive patients, the original maintenance treatment (eg. immunotherapy or immunotherapy combined with chemotherapy) will be continued.
  Interventions: Other: Standard Treatment
- Escalation Treatment (Experimental): For ctDNA-positive patients, escalated treatment will be administered.
  Interventions: Drug: Ivonescimab plus docetaxel

INTERVENTIONS:
Drug: Ivonescimab plus docetaxel — For ctDNA-positive patients, escalation treatment will be administrated
  1. Ivonescimab: Intravenous infusion (IV), 20 mg/kg, Day 1, every 3 weeks (Q3W);
  2. Docetaxel: IV, 75 mg/m², Day 1, Q3W (The investigator may adjust the chemotherapy dose and schedule based on the patient's tolerance during treatment.)
  All enrolled participants will continue treatment until one of the following occurs, whichever comes first:
  * The investigator determines that there is no longer clinical benefit (based on imaging assessments and clinical status)
  * Unacceptable toxicity
  * Completion of 24 months of treatment
  * Other discontinuation criteria specified in the protocol are met.
  Arms: Escalation Treatment
Other: Standard Treatment — For ctDNA-positive patients, continuing the original immunotherapy maintenance or immunotherapy combined with chemotherapy
  • In the event of clinical progression, consider switching to treatment with Ivonescimab plus docetaxel, administered every 3 weeks.
  Arms: Standard Treatment

SUMMARY:
The CR1STAL-Adaptive study is a randomized, open-label, phase II multicenter interventional trial designed to evaluate the safety and efficacy of Ivonescimab (PD-1/VEGF bispecific antibody) combined with docetaxel versus standard treatment in patients with advanced NSCLC who have achieved long-term benefit from first-line immune checkpoint inhibitors (ICIs), but are ctDNA-MRD positive. Building upon insights from previous CR1STAL study (NCT05198154), the CR1STAL-Adaptive study supports the development of precision-guided, adaptive treatment strategies to delay progression and improve outcomes in NSCLC patients with a long-term response to immunotherapy. It represents a step forward in integrating dynamic molecular monitoring with individualized intervention strategies in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent prior to any study-related procedures, be willing and able to complete the visits, treatment regimen, and laboratory tests specified in the schedule, and comply with other requirements of the study;
2. Aged ≥18 and ≤75 years old;
3. ECOG PS score 0-1;
4. Expected survival time ≥ 12 weeks;
5. Patients with stage IIIB-IIIC and IV non-small cell lung cancer confirmed by histology or cytology that cannot be treated locally (TNM lung cancer staging of the 9th edition of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification);
6. There must be no EGFR gene-sensitive mutation, ALK gene fusion or ROS1 gene fusion in non-squamous carcinoma
7. Immunotherapy combined with platinum-containing doublet chemotherapy as a first-line standard treatment regimen;
8. Non-PD with PFS at screening enrollment is 11 to 15 months;
9. According to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1), it is recommended to have at least one measurable lesion, but patients without measurable lesions can still be included in the group (primary tumor recurrence or new metastatic lesions are considered PD).

Participants with brain metastases who are asymptomatic or whose symptoms are stable after local treatment are allowed to enroll, as long as the participants meet the following conditions:

1. There are measurable lesions outside the central nervous system
2. No central nervous system symptoms or no worsening of symptoms for at least 2 weeks
3. No need for glucocorticoid treatment, or glucocorticoid treatment was discontinued within 7 days before the first dose, or the glucocorticoid dosage was stable and reduced to less than 10mg/day prednisone (or equivalent dose) within 7 days before the first dose.

10. Meet the following laboratory indicators (within 14 days before the first treatment):

1. Routine blood test: absolute neutrophil count ≥1.5×109/L; platelet count ≥100×109/L; hemoglobin content ≥9.0 g/dL (no blood transfusion or erythropoietin-dependent administration within 7 days).
2. Liver function: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); for patients with liver metastasis or confirmed/suspected Gilbert's syndrome, TBIL ≤3×ULN; in the absence of liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. For patients with liver metastasis, ALT or AST ≤5×ULN.
3. Renal function: serum creatinine (Cr) ≤ 1.5 times ULN or Cr clearance ≥ 50 mL/min (Cockcroft-Gault formula), and urine routine test results show urine protein (UPRO) <2+ or 24-hour urine protein quantification <1g.
4. Coagulation function: international normalized ratio (INR) ≤ 1.5 times ULN or partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; if the study participants are receiving anticoagulant therapy, as long as PT is within the range of the anticoagulant drug;
5. Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% 11. For female study participants of childbearing age, a urine or serum pregnancy test with a negative result should be performed within 3 days before the first dose of study drug (Day 1 of Cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-childbearing age are defined as women who have been postmenopausal for at least 1 year, or have undergone surgical sterilization or hysterectomy; if there is a risk of pregnancy, all study participants (whether male or female) must use contraceptive measures with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of study drug).

12. If an intact male study participant has sexual intercourse with a female partner of reproductive potential, the study participant must use effective contraception from screening until day 120 after the last dose. Whether to discontinue contraception after this time point should be discussed with the investigator.

Exclusion Criteria:

1. Concurrent participation in another interventional clinical study or receipt of another investigational drug, unless participating in an observational clinical study；
2. Systemic therapy with proprietary Chinese medicines with anti-tumor indications or immunomodulatory drugs (including thiopeptides, interferons, interleukins, except those used locally for the control of hydrothorax or ascites) within 2 weeks prior to the first dose；
3. No measurable lesions as defined by RECIST 1.1 due to prior radical treatment (e.g., surgery or radiotherapy)
4. Subjects who have received systemic antiangiogenic therapy;
5. Subjects who are enrolled in another clinical study at the same time, unless it is a non-interventional clinical study or the follow-up period of an interventional study (defined as the time between the first dose of this study and the last dose of the previous clinical study being more than 4 weeks or more than 5 half-lives of other study drugs, whichever is shorter);
6. During the screening period, imaging shows that the tumor surrounds important blood vessels or there is significant necrosis or cavity, and the investigator determines that entering the study will cause a risk of bleeding;
7. Imaging findings during the screening period show that the tumor invades important peripheral organs and blood vessels (such as the heart and pericardium, trachea, esophagus, aorta, superior vena cava, etc.) or there is a risk of developing esophagotracheal fistula or esophagopleural fistula;
8. Active autoimmune diseases requiring systemic treatment (such as treatment with disease-modifying drugs, corticosteroids, and immunosuppressants) within 2 years before the first dose (excluding irAEs caused by the use of PD-1/L1 inhibitors). Replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a systemic treatment;
9. A history of major diseases within 1 year before the first dose, specifically:

   * Unstable angina, myocardial infarction, congestive heart failure (NYHA classification ≥ Class 2) or vascular diseases (such as aortic aneurysm with a risk of rupture) that require hospitalization within 12 months before the first dose, or other cardiac damage that may affect the safety evaluation of the study drug (such as poorly controlled arrhythmia, myocardial ischemia, etc.);
   * Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh class B or more severe cirrhosis
   * Current hypertension with systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive therapy;
   * Hyperglycemia that cannot be controlled after treatment (fasting blood glucose > 10 mmol/L);
   * A history of esophageal and gastric varices, with severe ulcers and unresolved wounds, abdominal fistulas, intraabdominal abscesses, or acute gastrointestinal bleeding within 6 months before the first dose;
   * Any arterial thromboembolic events, venous thromboembolic events of grade 3 orabove as specified in NCI CTCAE 5.0, transient ischemic attacks, cerebrovascular accidents, hypertensive crises, or hypertensive encephalopathy that occurred within 6 months before the first dose;
   * Acute exacerbation of chronic obstructive pulmonary disease that occurred within 4 weeks before the first dose;
   * Active or prior history of inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea);
10. A history of gastrointestinal perforation and/or fistula, a history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), or extensive bowel resection (partial colon resection or extensive small bowel resection, with chronic diarrhea) within 6 months before the first dose;
11. Those who have received chest radiotherapy >30 Gy within 6 months before the first dose, non-chest radiotherapy >30 Gy within 4 weeks before the first dose, and palliative radiotherapy ≤ 30 Gy within 2 weeks before the first dose, and who have not recoveredfrom the toxicity and/or complications of these interventions to NCI-CTC AE ≤ grade 1 (excluding alopecia and fatigue). Palliative radiotherapy to control symptoms is allowed, but it must be completed at least 2 weeks before the first dose, and no additional radiotherapy is scheduled for the same lesion;
12. Those who have received live or live attenuated vaccines within 4 weeks before the first dose, or plan to receive live or live attenuated vaccines during the study period. The use of inactivated vaccines is allowed;
13. Severe infections within 4 weeks before the first dose, including but not limited to complications requiring hospitalization such as sepsis, or severe pneumonia; active infections that have received systemic anti-infective treatment within 2 weeks before the first dose (excluding antiviral treatment for hepatitis B or C);
14. Those with a history of severe bleeding tendencies or coagulation disorders; those with clinically significant bleeding symptoms within 4 weeks before the first dose, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or vomiting up ≥ 1 teaspoon of blood or small blood clots, or only coughing up blood without sputum; those with blood in the sputum are allowed to be enrolled), nasal bleeding (excluding epistaxis and bloody nasal discharge); those who have received continuous antiplatelet or anticoagulant therapy (except for preventive use of anticoagulants, such as the use of anticoagulants to maintain venous patency) within 14 days before the first dose;
15. Those who have undergone major surgery or experienced severe trauma within 4 weeks before the first dose, or have a major surgery planned within 4 weeks after the first dose (as determined by the investigator);
16. Presence of clinically uncontrolled pleural effusion or ascites (subjects may be recruited who do not require drainage of the effusion or who do not have a significant increase in the effusion after 3 days of cessation of drainage)
17. Previous history of non-infectious pneumonia requiring systemic glucocorticoid treatment or current interstitial lung disease;
18. Those with a history of immunodeficiency; those with positive HIV antibody tests;
19. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
20. Subjects with untreated active hepatitis B (HBsAg positive and HBV-DNA > 1000 copies/mL (200 IU/mL) or above the lower limit of detection, whichever is higher), for subjects with hepatitis B who are required to receive anti-hepatitis B virus treatment during the study treatment period; subjects with active hepatitis C subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
21. Known presence of active pulmonary tuberculosis (TB);
22. Known active syphilis infection;
23. Known allergy to any component of any study drug; a known history of severe hypersensitivity to other monoclonal antibodies
24. Those with a history of immunodeficienc; those who are currently receiving long-term systemic corticosteroids or other immunosuppressants;
25. A known history of mental illness, drug abuse, alcohol or drug addiction;
26. The toxicity of previous anti-tumor therapy has not been relieved, which is defined as the toxicity has not returned to grade 1 or below specified in NCI CTCAE 5.0, or the level specified in the inclusion/exclusion criteria, except for alopecia and fatigue;
27. Known symptomatic CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may be enrolled in the trial if they are clinically stable (no evidence of imaging progression for at least 4 weeks prior to the first dose of the experimental treatment, no evidence of new brain metastases or increase in size of pre-existing brain metastases as confirmed by repeat imaging) and do not require steroid therapy for at least 14 days prior to the first dose of the experimental treatment. This exception does not include carcinomatous meningitis, which should be excluded regardless of whether it is clinically stable.
28. History of other primary malignancies within 5 years, except：

    * malignancies that have been in complete remission for at least 2 years prior to enrolment and for which no other treatment was required during the study period.
    * adequately treated non-melanoma skin cancer or malignant nevus with no evidence of disease recurrence.
    * adequately treated carcinoma in situ without evidence of disease recurrence
29. Subjects who are pregnant or breastfeeding or plan to breastfeed during the study;
30. Other acute or chronic illnesses, psychiatric disorders, or abnormal laboratory test values that could increase the risks associated with study participation or study drug administration or interfere with the interpretation of study results and, in the investigator's judgment, render the patient ineligible for participation in the study.
31. Uncontrolled metabolic disorders, or local or systemic diseases due to non-malignant tumors, or diseases or symptoms secondary to the tumor, which may lead to higher medical risk and/or uncertainty in survival assessment, or diseases that the investigator considers unsuitable for enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in ctDNA-Positive Population | 3 years
  The time from detection of ctDNA-MRD positivity to disease progression or death.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) in the Overall Population | 3 years
  The time from enrollment to disease progression or death in the entire population (including both ctDNA-positive and ctDNA-negative participants).
Overall Survival (OS) | 5 years
  The time from study enrollment to death from any cause.
Adverse Events (AEs) | 3 years
  During the study period and follow-up, the severity of adverse events will be graded based on NCI CTCAE version 5.0. Safety evaluation indicators include:
  * The type, incidence, severity, and relationship to the study drug of all AEs, treatment-emergent AEs (TEAEs), serious AEs (SAEs), and immune-related AEs (irAEs);
  * The number and proportion of participants who discontinue treatment due to the above adverse events;
  * Changes in vital signs, physical examination findings, and laboratory test results before, during, and after the study treatment.
ctDNA Clearance | 3 years
  ctDNA clearance rate at Cycle 3 Day 1 (C3D1) after escalated treatment.
Objective Response Rate (ORR) | 3 years
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR).
  * DCR is defined as the proportion of participants achieving CR, PR, or stable disease (SD).
  * ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | 3 years
  DCR is defined as the proportion of participants achieving CR, PR, or stable disease (SD).
Quality of Life (QoL) | 3 years
  Quality of life (QoL) is assessed longitude by EORTC QLQ-C30 (version.3). The EORTC QLQ-C30 is composed of 9 multi-item scales: 5 functioning scales (physical, role, cognitive, emotional, and social), a global QOL scale, and 3 symptom scales (fatigue, pain, and nausea/vomiting). All scales and single items are linearly transformed to an 0-100 scale. A higher score represents a better level of functioning.

OTHER OUTCOMES:
Biomarkers | 3 years
  The ctDNA dynamics when patients receive the escalation treatment.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Hunan Cancer Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - The First Hospital of Changsha, Changsha
  - Army Medical Center (Daping Hospital), Chongqicun
  - Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong
  - The First Affiliated Hospital of Guangxi Medical University, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang